CLINICAL TRIAL: NCT02005653
Title: Alternate Chemotherapy Regimens for the Clearance of W.Bancrofti Infection: Double Blind Randomised Clinical Trial (RCT) to Study the Efficacy of Different Co-administration and Sequential Administration
Brief Title: Alternate Chemotherapy Regimens for the Clearance of W.Bancrofti Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Lourduraj John De Britto, Scientist-E (Medical), Indian Council of Medical Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM0603-CEC-VCRC
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Filarial; Infestation
Keywords: Lymphatic filariasis; W. bancrofti; DEC; Albendazole; Doxycycline
MeSH Terms: conditions — Parasitic Diseases; Elephantiasis, Filarial | interventions — Diethylcarbamazine; Albendazole; Albumins; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DEC + ALB sequential (Experimental): Diethylcarbamazine 300 mg tablet and albendazole 400 mg tablet at 30 days post treatment sequentially
  Interventions: Drug: Diethylcarbamazine; Drug: Albendazole
- DEC + ALB co-admin (Experimental): Diethylcarbamazine 300 mg tablet and albendazole 400 mg tablet per day given orally as single dose for 12 days
  Interventions: Drug: Diethylcarbamazine; Drug: Albendazole
- DEC + DOXY co-admin (Experimental): Diethylcarbamazine 300 mg tablet and Doxycycline 100 mg per day given orally as single dose for 12 days
  Interventions: Drug: Diethylcarbamazine; Drug: Doxycycline
- Diethylcarbamazine (DEC) (Active Comparator): Diethylcarbamazine 300 mg tablet as single dose orally per day for 12 days
  Interventions: Drug: Diethylcarbamazine

INTERVENTIONS:
Drug: Diethylcarbamazine — Diethylcarbamazine 300 mg tablet as single dose per day for 12 days
  Other Names: DEC
Drug: Albendazole — Experimental
  Other Names: Alb
  Arms: DEC + ALB co-admin; DEC + ALB sequential
Drug: Doxycycline — Experimental
  Other Names: Doxy
  Arms: DEC + DOXY co-admin

SUMMARY:
Diethylcarbamazine (DEC) essentially a micro-filaricidal drug is given for 12 days as standard treatment for the clearance of W. bancrofti infection. It takes about one year for the individuals to completely clear the microfilaria from the blood. It takes another two to four years to clear the antigen. The aim of the present study is to shorten the time taken for clearing the Mf and antigen from the blood either by co-administration or sequential administration of a macrofilaricidal drug, Albendazole or doxycycline. This study is a randomized, double blind, controlled clinical trial to study the efficacy of these drug combinations in complete clearance the Mf and antigen from the blood in shorter span of 180 days and 365 days respectively.

DETAILED DESCRIPTION:
Purpose:

Lymphatic dwelling parasite W. bancrofti is the most common cause of secondary lymphoedema. Till today, there is no effective treatment protocol for the complete clearance of W. bancrofti infection, in a short duration of time.

Methods:

The investigators conducted a double blind RCT under field conditions recruiting 146 asymptomatic W. bancrofti infected individuals. Participants were randomly assigned one of the four regimens for 12 days, DEC 300 mg + Doxycycline 100 mg co-administration or DEC 300 mg + Albendazole 400 mg co-administration or DEC 300 mg + Albendazole 400 mg sequential administration or control regimen DEC 300 mg. Participants were followed up at 13, 26 and 52 weeks post-treatment for the clearance of infection.

ELIGIBILITY:
Inclusion Criteria:

* Residing in or around Pondicherry and adjoining Tamilnadu areas
* Night blood microfilaria counts > 10 mf/ml by membrane filtration
* No history of treatment for filarial infection for the last two years at least
* Willing for home visits by the staff of the center
* Willing to give written informed consent

Exclusion Criteria:

* Body weight less than 30 kg
* Hepatic or renal disease as evidenced by clinical or biochemical abnormalities. - concurrent illness like hypertension, diabetes mellitus, cardiac conditions and epilepsy requiring chronic medication
* Psychiatric illness
* Patients under tetracycline or doxycycline therapy
* History of de-worming by albendazole or other anti-helminthic during last one year
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
complete clearance of mf in 80% of the infected | At 13th week (91 days) post therapy

SECONDARY OUTCOMES:
Complete clearance Mf and complete clearance of antigen from the infected | 26 and 52 weeks post therapy
  a)Complete clearance of Mf by 26 weeks (180 days) post therapy. b) Complete clearance of antigen by 52 weeks (365days) post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lourduraj J De Britto, M.D, Principal Investigator — Vector Control Research Centre, Indian Council of Medical Research, Pondicherry
Locations (1):
- Vector Control Research Centre, Puducherry, Puducherry, India

REFERENCES:
- [Derived] De Britto RL, Vanamail P, Sankari T, Vijayalakshmi G, Das LK, Pani SP. Enhanced efficacy of sequential administration of Albendazole for the clearance of Wuchereria bancrofti infection: Double blind RCT. Trop Biomed. 2015 Jun;32(2):198-209. PMID 26691247